CLINICAL TRIAL: NCT06589141
Title: Comparison Between Metformin and Glyburide in the Management of Gestational Diabetes: a Randomized Controlled Trial (GDM-MERGE Trial)
Brief Title: Comparison Between Metformin and Glyburide in the Management of Gestational Diabetes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Collaborators: Middle-Eastern College of Obstetricians and Gynecologists (Other)
Responsible Party: Principal Investigator, Sherif Abdelkarim Mohammed Shazly, Senior clinical fellow, Middle-Eastern College of Obstetricians and Gynecologists
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: GDM-MERGE trial
Record Dates: First submitted 2024-08-26; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Gestational Diabetes Mellitus in Pregnancy
Keywords: Metformin and Glyburide
MeSH Terms: interventions — Metformin; Tablets; Glyburide

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metformin (Experimental): Metformin (500 to 2000 mg orally)
  Interventions: Drug: MetFORMIN 500 Mg Oral Tablet
- Glyburide (Experimental): Glyburide (2.5 mg to 20 mg orally)
  Interventions: Drug: GlyBURIDE 2.5 MG Oral Tablet

INTERVENTIONS:
Drug: MetFORMIN 500 Mg Oral Tablet — Metformin (500 to 2000 mg orally)
  Arms: Metformin
Drug: GlyBURIDE 2.5 MG Oral Tablet — Glyburide (2.5 mg to 20 mg orally)
  Arms: Glyburide

SUMMARY:
This study aims to compare the maternal, fetal, and neonatal outcomes associated with the use of metformin versus glyburide for managing gestational diabetes.

The objective is to assess the safety and effectiveness profiles of both medications as potential alternatives to initiating insulin therapy.

DETAILED DESCRIPTION:
Primary Outcome: treatment failure is defined as the initiation of insulin due to failure of glycemic control (more than 10% of high values using 4-point glucose checks) or side effects.

Secondary Outcomes:

Maternal:

* Percentage of fasting and postprandial glucose levels within target levels after initiation of treatment
* Incidence of maternal hypoglycemia
* Reported maternal side effects
* Maternal weight gain
* Preterm delivery
* Development of pregnancy-induced hypertension
* Labor dystocia.
* Instrumental delivery and its indication (fetal compromise, delay in progress, or maternal exhaustion)
* Mode of delivery
* Incidence of third and fourth perineal tear

Fetal and neonatal:

* Fetal large for gestational age
* Intrauterine fetal death
* Newborn weight
* Gestational age at delivery
* Neonatal birth injuries
* Stillbirth and neonatal death
* Apgar score at 1 minute

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women over 18 years old.
* Gestational age between 24 - 28 weeks.
* New diagnosis of gestational diabetes mellitus using a 2-hour glucose tolerance test.
* Medical therapy is indicated to control blood glucose following the failure of diet and lifestyle changes to solely achieve glycemic control (A2GDM).

Exclusion Criteria:

Patients with pre-gestational diabetes.

* First trimester fasting blood glucose ≥105 mg/dl or HbA1c > 6.4%.
* Major fetal anomalies.
* Intrauterine growth restriction (IUGR) before 24 weeks.
* Abnormal renal or liver function.
* Contraindications to metformin or glyburide.
* Medical treatment declined by the patient.
* Direct indication to commence insulin (initial fasting blood glucose >= 7 mmol/l or 126 mg/dl or >= 6 mmol/l or 108 mg/dl with macrosomia or polyhydramnios).
* Significant medical co-morbidities requiring continuous medical treatment in pregnancy.
* Non-compliance to blood glucose self-monitoring (missing 50% or more of total readings)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 180 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Treatment failure | From 28 weeks till 41 weeks of pregnancy
  Initiation of insulin due to failure of glycemic control (more than 10% of high values using 4-point glucose checks) or side effects

SECONDARY OUTCOMES:
Incidence of maternal hypoglycemia | From 28 weeks till 41 weeks of pregnancy
  Incidence of blood glucose levels below 4 mmol/L during the period of treatment
Significant side effects | From 28 weeks till 41 weeks of pregnancy
  Incidence of maternal significant side effects requiring cessation of treatment (gastrointestinal side effects)
Fetal macrosomia (large for gestational age) | 32 weeks of gestation to onset of labour
  Incidence of fetuses growing above the 90th percentile on third ultrasound scan using customised growth chart

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ye W, Luo C, Huang J, Li C, Liu Z, Liu F. Gestational diabetes mellitus and adverse pregnancy outcomes: systematic review and meta-analysis. BMJ. 2022 May 25;377:e067946. doi: 10.1136/bmj-2021-067946. PMID 35613728
- [Background] Silva JC, Fachin DR, Coral ML, Bertini AM. Perinatal impact of the use of metformin and glyburide for the treatment of gestational diabetes mellitus. J Perinat Med. 2012 Jan 10;40(3):225-8. doi: 10.1515/jpm-2011-0175. PMID 22505499
- [Background] Shuster DL, Shireman LM, Ma X, Shen DD, Flood Nichols SK, Ahmed MS, Clark S, Caritis S, Venkataramanan R, Haas DM, Quinney SK, Haneline LS, Tita AT, Manuck TA, Thummel KE, Brown LM, Ren Z, Brown Z, Easterling TR, Hebert MF. Pharmacodynamics of Glyburide, Metformin, and Glyburide/Metformin Combination Therapy in the Treatment of Gestational Diabetes Mellitus. Clin Pharmacol Ther. 2020 Jun;107(6):1362-1372. doi: 10.1002/cpt.1749. Epub 2020 Jan 25. PMID 31869430
- [Background] Oliveira MM, Andrade KFO, Lima GHS, Rocha TC. Metformin versus glyburide in treatment and control of gestational diabetes mellitus: a systematic review with meta-analysis. Einstein (Sao Paulo). 2022 Feb 16;20:eRW6155. doi: 10.31744/einstein_journal/2022RW6155. eCollection 2022. PMID 35195193